CLINICAL TRIAL: NCT03498495
Title: Kids With mTBI Get SMART: Development and Pilot Trial of a Web-Based Self-Monitoring Activity-Restriction and Relaxation Training Program
Brief Title: Web-Based Self-Monitoring Activity-Restriction and Relaxation Training Program for Kids With Mild Traumatic Brain Injury
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIN001--SMART
Record Dates: First submitted 2018-04-04; First posted 2018-04-13 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Brain Injury Traumatic Mild
MeSH Terms: conditions — Brain Concussion | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART Intervention (Experimental)
  Interventions: Behavioral: Self-Monitoring Activity-restriction and Relaxation Training (SMART)
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Self-Monitoring Activity-restriction and Relaxation Training (SMART) — SMART integrates real-time self-monitoring of symptoms and activities with interactive modules designed to increase self-efficacy through psychoeducation and training in problem solving/problem-focused coping strategies.
  Arms: SMART Intervention

SUMMARY:
SMART is an interactive web-based program that will allow youth with mild traumatic brain injuries (mTBI) to monitor their symptoms and receive education on problem-solving and coping strategies. This study will evaluate the effectiveness of SMART as a means of improving symptom-management, coping skills, and general well-being during recovery from mTBI. Half of participants will receive the SMART intervention, while half will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* 11-18 years old
* Sustained mTBI within the past week

Exclusion Criteria:

* Patient and/or family do not speak and read English
* Patient and/or family do not have Internet access
* Patient experiencing more severe brain injury (Glasgow coma score <13)
* Patient with more than one moderate extracranial injury
* Patients with non-mTBI reasons for altered mental status
* Patients with severe pre-existing neurologic or cognitive disorders or other disorders that may impair ability to participate in the intervention.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in quality of life, as measured by the Pediatric Quality of Life Inventory (PedsQL) | From baseline to 4 weeks post-injury
  The PedsQL includes 23 items measuring physical, emotional, social, and school functioning.

SECONDARY OUTCOMES:
Change in coping strategies, as measured by the Coping Strategies Inventory (CSI-S: Short Form) | From baseline to 4 weeks post-injury
  The CSI-S is a coping styles measure and has been used with other pediatric TBI samples. Adolescents rate how much they agree with 32-statements regarding different ways of coping with difficult situations on a 5-point Likert scale. Responses are then grouped into primary subscales reflecting eight different coping strategies (e.g., problem-solving, problem avoidance, social withdrawal, etc.).
Change in self-efficacy for symptom management, as measured by the Self-Efficacy Scale (S-eS) | From baseline to 4 weeks post-injury
  This 2-item measure will be developed by the research team based on Bandura's self-efficacy theory. Adolescents will rate their level of confidence that they are able to maintain a plan to manage their symptoms each week
Change in general functioning, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) | From baseline to 4 weeks post-injury
  PROMIS collects data from the adolescent participant and the parent about the impact a condition has on the adolescent's functioning.
Change in health and behavioral symptoms, as measured by the Health and Behavior Inventory (HBI) | From baseline to 4 weeks post-injury
  The HBI is a 20-item questionnaire which includes a variety of cognitive, somatic, emotional, and behavioral symptoms requiring parents and adolescents to rate the frequency of occurrence of each symptom over the past week on a 4-point scale, ranging from "never" to "often."

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Babcock, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wade SL, Sidol C, Babcock L, Schmidt M, Kurowski B, Cassedy A, Zhang N. Findings from a Randomized Controlled Trial of SMART: An EHealth Intervention for Mild Traumatic Brain Injury. J Pediatr Psychol. 2023 Mar 20;48(3):241-253. doi: 10.1093/jpepsy/jsac086. PMID 36565462

DOCUMENTS (1):
  • Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT03498495/ICF_000.pdf